CLINICAL TRIAL: NCT06790511
Title: Clinical Performance of Bioactive Highly Filled Injectable Flowable Composite for Direct Posterior Occlusal Conservative Restorations Using FDI Criteria: Two Year Randomized Clinical Trial
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Sherif, Ass. Lectuerer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mohamed Sherif PHD
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: highly filled injectable flowable composite
- Intervention (Experimental)
  Interventions: Other: bioactive highly filled injectable flowable composite

INTERVENTIONS:
Other: bioactive highly filled injectable flowable composite — bioactive highly filled injectable flowable composite
  Other Names: Shofou Flow Plus X
  Arms: Intervention
Other: highly filled injectable flowable composite — highly filled injectable flowable composite
  Other Names: GC G-ænial Universal Flo
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate Clinical Performance of bioactive highly filled injectable flowable composite for direct posterior occlusal conservative restorations using FDI Criteria

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria: patient age range from 16-45 years, with a premolar indicated for extraction, patients required at least a couple of Class I restorations. The patient should have good general health.

-

Exclusion Criteria:Where the exclusion criteria will be: poor oral hygiene, sever or chronic periodontal disease or bruxism, severe tooth sensitivity, non-vital or fracture or cracked teeth, defective restorations or bleaching procedures during the last 6 months, pregnancy, and/or lactation, and allergy to the main components of the products to be used in the study.

-

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of caries | 24 Months
  Restorations will be assessed for recurrence of caries by visual examination, short air drying

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol